CLINICAL TRIAL: NCT07378150
Title: The Effect of Clay Therapy on Functional Improvement and Individual and Social Performance in Schizophrenic Patients
Brief Title: Clay Therapy in Schizophrenia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Esra Karabulut, Lecturer, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSHU-SBF-EK-01
Record Dates: First submitted 2025-08-26; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia and Related Disorders
Keywords: schizophrenia; clay therapy; Functional Recovery; Individual and Social Performance; art therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Two groups with a conventional therapy control group
Who Masked: Participant, Outcomes Assessor
Masking Description: While the conventional treatment group continues to receive routine treatment, the experimental group will receive clay therapy sessions in addition to treatment, and the outcome assessments will be conducted by a researcher who is unaware of the group distribution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clay therapy group (Experimental): The experimental group will receive clay therapy sessions in addition to routine therapies.
  Interventions: Other: Clay therapy
- Routine treatment group (No Intervention): Routine therapies will continue to be administered to the control group, but clay therapy will not be administered.

INTERVENTIONS:
Other: Clay therapy — Experimental: Clay therapy group
  Arms: Clay therapy group

SUMMARY:
In recent years, art therapies have been discussed for their positive effects on mental disorders. One such therapy, clay therapy, is being studied to examine its effect on the functional recovery and individual and social performance of schizophrenia patients undergoing pharmacological treatment.

DETAILED DESCRIPTION:
Schizophrenia is a chronic illness that can manifest in various forms, ranging from symptoms such as delusions and hallucinations to functional impairments, and is often characterised by relapses.

The care of people with schizophrenia concerns all sectors of society, including families, healthcare professionals, and organisations providing psychosocial support. The treatment of schizophrenia is of great importance due to its potential for early onset and its status as one of the most common psychiatric disorders leading to functional impairment.

While pharmacological treatments support a large part of the treatment process, the effect of art therapy on preventing disability and treatment compliance and disease awareness is the subject of current studies. Clay therapy, a component of art therapy, has been used in the treatment of psychiatric disorders, especially in recent years. Studies have highlighted the therapeutic aspects of clay. When examining the therapeutic properties of clay, it is seen to provide benefits in the following areas:

* Facilitating the expression of emotions,
* Bringing unconscious material to the surface,
* Facilitating rich and deep expression,
* Facilitating verbal communication,
* Concretisation and symbolisation. This study aims to examine the effect of clay therapy on the functional recovery and individual and social performance of schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with schizophrenia,
* Being aged 18 or over,
* Having completed at least primary school education,
* Having achieved treatment compliance,
* Currently undergoing pharmacological treatment,
* Being in remission,
* Having attended the Community Mental Health Centre regularly over the past year,
* Having agreed to participate in the study
* Scoring 20 points or higher on the Mini Mental State Examination

Exclusion Criteria:

* Being under 18 years of age,
* Not having an education,
* Not having a diagnosis of schizophrenia,
* Not adhering to treatment,
* Not taking pharmacological treatment regularly,
* Being in an acute attack/active phase,
* Lacking insight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Functional Recovery Scale for Schizophrenia Patients | 12 weeks
  This is a 5-point Likert-type scale consisting of 19 items that assesses improvements in functionality independent of the symptoms of the disease. Level 1 (absent) indicates the lowest level of improvement, while Level 5 (present to a high degree) corresponds to the 'ideal' level of function. Level 2 (partially present), Level 3 (sufficiently present) and Level 4 (almost completely present) are also included. When two levels are between, the lower level is selected. The maximum score that can be obtained from the scale is 95, and the minimum score is 19. The scale, which consists of subscales for daily living skills, social functioning, and health and treatment, measures functional improvement in three separate areas.

SECONDARY OUTCOMES:
Individual and Social Performance Scale | 12 weeks
  This scale, scored from 1 to 100, is conducted in three stages. In the first stage, the level of functionality is determined through a sequential assessment across four dimensions: socially beneficial activities, individual and social relationships, self-care, and disruptive and aggressive behaviours. After each dimension is assessed, it is scored between 0 and 10 points based on the degree of impairment in that dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Kutahya Health Sciences University, Kütahya, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Utas-Akhan, L.., Avci, D., Basak, I. 2024. "Art Therapy as a nursing intervention for individuals with schizophrenia", Journal of Psychosocial Nursing and Mental Health Services, 62(5), 29-38. https://doi.org/10.3928/02793695-20231025-02
- [Background] Cataldas, S. K., Eren, N., Üstün, N., Ofluoğlu, F., Ayhan, C. H. 2025. "Effects of art therapy on quality of life and social functioning in individuals with schizophrenia", Journal of Psychosocial Nursing and Mental Health Services, 0(0), 1-7. https://doi.org/10.3928/02793695-20250107-02
- [Background] Ursuliak Z, Hughes J, Crocker CE, MacKenzie A, Tibbo PG. Claymation art therapy in early phase psychosis: A qualitative study to explore participants' experiences with the program and identify outcome effects. Early Interv Psychiatry. 2020 Dec;14(6):698-704. doi: 10.1111/eip.12896. Epub 2019 Nov 6. PMID 31692270
- [Background] Taksal A, Sudhir PM, Janakiprasad KK, Viswanath D, Thirthalli J. Feasibility and effectiveness of the Integrated Psychological Therapy (IPT) in patients with schizophrenia: a preliminary investigation from India. Asian J Psychiatr. 2015 Oct;17:78-84. doi: 10.1016/j.ajp.2015.06.013. Epub 2015 Jul 30. PMID 26277224